CLINICAL TRIAL: NCT00969306
Title: Chloroquine as an Anti-autophagy Drug in Stage IV Small Cell Lung Cancer (SCLC) Patients: A Phase 1 Trial
Brief Title: Chloroquine as an Anti-Autophagy Drug in Stage IV Small Cell Lung Cancer (SCLC) Patients
Acronym: Chloroquine IV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chloroquine IV
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Chloroquine

ARMS (1):
- Chloroquine (Active Comparator): Patients receive Chloroquine
  Interventions: Drug: Chloroquine, A-CQ 100

INTERVENTIONS:
Drug: Chloroquine, A-CQ 100 — Administration:
  * Orally
  * Timing: Once daily
  * Tablets of 100 mg
  * During or after meals
  * In case of missed dose: intake of the missed dose is still possible up until 12 hours before the next dose.
  * Patients should always note date and time of intake on the chloroquine monitoring form.

SUMMARY:
Chloroquine might very well be able to increase overall survival in small cell lung cancer by sensitizing cells resistant to chemotherapy and radiotherapy.

DETAILED DESCRIPTION:
Tumor hypoxia is a well-known factor negatively influencing outcome in many solid tumors, including small cell lung cancer. Hypoxic cells are more radio-resistant, more chemo-resistant and more prone to develop distant metastases than normoxic cells.

One of the mechanisms responsible for survival of these therapy-resistant hypoxic cells is (macro-)autophagy: a phenomenon in which cells provide themselves with energy (ATP) by digesting their own cell-organelles. Chloroquine is a potent blocker of autophagy and has been demonstrated in a lab setting to dramatically enhance tumor response to radiotherapy, chemotherapy and even anti-hormonal therapy.

Thus, chloroquine might very well be able to increase overall survival in small cell lung cancer by sensitizing cells resistant to chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ''extensive disease'' (Stage T0-4 N0-3 M1) small cell lung cancer
* At least one measurable disease site, defined as lesion of ≥ 1 cm unidimensionally on CT-scan.
* WHO performance status 0-2
* Absolute neutrophil count at least 1800/µl and platelets at least 100000/µl and hemoglobin at least 6.2 mmol/l.
* Calculated creatinine clearance at least 60 ml/min
* Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution (in case of liver metastases ≤ 5 x ULN for the institution)
* No previous platinum chemotherapy or topo-isomerase-inhibitors for SCLC.
* Life expectancy more than 6 months
* Willing and able to comply with the study prescriptions
* 18 years or older
* Not pregnant or breast feeding and willing to take adequate contraceptive measures during the study
* Ability to give and having given written informed consent before patient registration
* No mixed pathology, e.g. non-small cell plus small cell cancer
* No recent (< 3 months) severe cardiac disease (NYHA class >1) (congestive heart failure, infarction)
* No history of cardiac arrythmia (multifocal premature ventricular contractions, uncontrolled atrial fibrillation, bigeminy, trigeminy, ventricular tachycardia) which is symptomatic and requiring treatment (CTC AE 4.0), or asymptomatic sustained ventricular tachycardia. Asymptomatic atrial fibrillation controlled on medication is allowed.
* No cardiac conduction disturbances or medication potentially causing them:
* QTc interval prolongation with other medications that required discontinuation of the treatment
* Congenital long QT-syndrome or unexplained sudden death of first degree relative under 40 years of age
* QTc interval > 480 msec (note: when this is the case on screening ECG, the ECG may be repeated twice. If the average QT-interval of these 3 measurements remains below 480 msec, patient is eligible)
* Patients on medication potentially prolongating the QT-interval are excluded if the QT-interval is > 460 msec (Appendix, table 2).
* Medication that might cause QT-prolongation or Torsades de pointes tachycardia is not allowed (Appendix, Table 1). Drugs with a risk of prolongating the QT-interval that cannot be discontinued are allowed, however, under close monitoring by the treating physician (Appendix, table 2).
* No uncontrolled infectious disease
* No other active malignancy
* No major surgery (excluding diagnostic procedures like e.g., mediastinoscopy) in previous 4 weeks
* No treatment with investigational drugs in 4 weeks prior to or during this study
* No chronic systemic immune therapy
* No known G6PD deficiency

Exclusion Criteria:

* The opposite of the above

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity of adding chloroquine in escalating doses in SCLC patients: to standard dose cisplatin-etoposide in extensive disease SCLC; to standard dose concurrent radiotherapy and cisplatin-etoposide in limited disease SCLC | 6 years

SECONDARY OUTCOMES:
Tumor response (according to RECIST) | 6 years
Overall survival | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, DM, PhD, Principal Investigator — Maastricht Radiation Oncology
Locations (4):
- Netherlands (4):
  - NKI/AvL, Amsterdam
  - VU Medical Center, Amsterdam
  - Maastricht Radiation Oncology, Maastricht
  - Maastricht University Medical Center, Maastricht